CLINICAL TRIAL: NCT04125862
Title: Elucidating Mechanisms of Pain in Adolescent and Adult Fibrous Dysplasia Patients
Brief Title: Pain in Fibrous Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jaymin Upadhyay, Assistant Professor, BCH, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P00030755
Record Dates: First submitted 2019-08-12; First posted 2019-10-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Fibrous Dysplasia/McCune-Albright Syndrome
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic

STUDY DESIGN:
Intervention Model Description: 2 parallel cohorts (FD/MAS patients and matched, healthy controls)
Who Masked: Participant
Masking Description: Individual performing data analyses will be blinded to whether dataset corresponds to FD/MAS patient or matched healthy control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fibrous Dysplasia/McCune-Albright Syndrome (Other): 20, Fibrous Dysplasia/McCune-Albright Syndrome Patients with or without pain
  Interventions: Diagnostic Test: MRI-based Neuroimaging; Diagnostic Test: Non-contrast MRI; Diagnostic Test: 18F-FDG-PET/CT; Diagnostic Test: 18F-NaF-PET/CT
- Healthy Controls (Other): 20, matched healthy controls
  Interventions: Diagnostic Test: MRI-based Neuroimaging

INTERVENTIONS:
Diagnostic Test: MRI-based Neuroimaging — During evoked pain fMRI, noxious pressure and heat stimuli will be applied in the two anatomical sites noted above. During fMRI data acquisition, a total of 5 pressure stimulations and 5 heat stimulations will be delivered. Both types of pain stimuli will be applied in a 36/17-sec off/on cycle. The off-condition will correspond to a baseline temperature of 35C and the on condition will match the subject-specific and site-specific 7/10 pressure and heat pain thresholds defined during QST procedures. VAS pain ratings associated with evoked pain stimulation will be collected at the end of each scan. The investigators will also explore the structural properties of the CNS by implementing high-resolution anatomical MRI (gray matter volumes) and diffusion tensor imaging (white matter pathway integrity). All CNS imaging will take approximately 50-60 minutes to complete
Diagnostic Test: Non-contrast MRI — Musculoskeletal imaging of the affected lower extremity. Patients will be allowed to watch a movie during data acquisition. The following MRI procedures will be completed in order to identify soft tissue lesions in active or painful regions. Fast spin echo (FSE) T2 fat saturated, T1 weighted MRI, FSE proton density MRI, Short-TI Inversion Recovery (STIR), Diffusion weighted MRI (DW-MRI) and 3D Double Echo Steady State (DESS) will be collected. All musculoskeletal MRI will take approximately 30 minutes to complete.
  Arms: Fibrous Dysplasia/McCune-Albright Syndrome
Diagnostic Test: 18F-FDG-PET/CT — Data will be collected 30 min after the intravenous administration of 18F-FDG with an expected average dose of approximately 200 MBq. CT data will be collected at a low-dose to minimize radiation exposure. Patients will be positioned supine head-first with arms on the side. The investigators project whole body data to be collected, but in some cases, the field of view may be limited to the patient's skull to below the knees. The data acquisition period is expected to last between 15-30 minutes and total radiation dose will be ~3-4 mSv.
  Arms: Fibrous Dysplasia/McCune-Albright Syndrome
Diagnostic Test: 18F-NaF-PET/CT — Data will be collected 30 min after the intravenous administration of 18F-NaF with an expected average dose of approximately 200 MBq. CT data will be collected at a low-dose to minimize radiation exposure. Patients will be positioned supine head-first with arms on the side. The investigators project whole body data to be collected, but in some cases, the field of view may be limited to the patient's skull to below the knees. The data acquisition period is expected to last between 15-30 minutes and total radiation dose will be ~3-4 mSv.
  Arms: Fibrous Dysplasia/McCune-Albright Syndrome

SUMMARY:
Pain remains a common and frequently debilitating symptom, particularly during adulthood of Fibrous Dysplasia/McCune-Albright Syndrome (FD/MAS). For many FD/MAS patients, the amount of pain perceived is not commensurate with the level of detectable musculoskeletal pathology. Using a combination of clinical and biological assessments, this investigation aims to understand what drives pain in FD/MAS.

DETAILED DESCRIPTION:
In Fibrous Dysplasia/McCune-Albright Syndrome (FD/MAS), healthy bone tissue and marrow is replaced with pre-osteoblastic, fibrous tissue, yielding skeletal deformities and an increased propensity towards fracture, musculoskeletal weakness and bone pain. Despite the frequent use of pharmacological and non-pharmacological analgesic strategies, pain in FD remains common and frequently debilitating, particularly during adulthood. Moreover, for many patients there is a discordance between perceived pain levels and detectable musculoskeletal pathology. To elucidate the mechanism underlying pain in FD/MAS patients, investigators at the National Institute of Dental and Craniofacial Research (NIDCR), National Center for Complementary and Integrative Heath (NCCIH) and Boston Children's Hospital (BCH) aim to probe three inter-related domains that are projected to underlie pain experience(s) in FD/MAS patients. These include (i.) the presence of maladaptive central nervous system processes that amplify afferent pain or somatosensory signals, and also facilitate persistent pain; (ii.) aberrant interplay between neurological and musculoskeletal systems; (iii.) a mental health status shaped by the overall burden of living with FD and (iv.) the influence of childhood, FD-related complications on adulthood pain phenotypes. To investigate these four domains hypothesized to underlie FD pain as well as inform on the disconnect between pain and FD disease burden, the investigators will employ methods that complement routine clinical evaluation and diagnostic tests (i.e., 18F-NaF PET/CT or 18F-FDG PET/CT) such as neuroimaging, musculoskeletal MRI and such as neuroimaging, musculoskeletal MRI and assessment of inflammatory and pain mediator expression in blood samples.

ELIGIBILITY:
Inclusion Criteria (FD/MAS patients):

* Male and Female subjects
* 10-45 years of age
* English Speaking ability sufficient to comprehend consent (with parental assistance if minor)
* Diagnosis of Fibrous Dysplasia

Exclusion Criteria for patients:

* Younger than 10 or older than 45 years old
* Weight > 285 lbs (weight limit of the MRI table and < 36lbs)
* Surgery leaving implanted material
* Contraindications to MRI scanning and PET scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia, previous significant research related exposure to ionizing radiation)

Exclusion Criteria for healthy controls:

Same as for the patients, with the addition of the following:

• Use of recreational or illicit drugs History of chronic pain

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
% signal difference in BOLD signal | 50-60 Minutes
  • % signal difference within striatal and limbic network structures during evoked-heat pain fMRI between FD/MAS patients with pain, FD/MAS patients without pain and matched, healthy volunteers.

SECONDARY OUTCOMES:
Numerical clinical pain rating score | 8 weeks
  • Numerical clinical pain rating score (NPRS, 0-10 scale) at weeks 0, 1, 4 and 8.

OTHER OUTCOMES:
18F-FDG or 18F-NaF uptake in FD lesion site | 15-30 Minutes
  18F-FDG or 18F-NaF Standard uptake value ratio in FD lesion site

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A two-way material transfer agreement has been executed between collaborating parties (Boston Children's Hospital and NIH)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual data will start to become available 12/2019 and last for 1.5 years.
Access Criteria: A two-way material transfer agreement